CLINICAL TRIAL: NCT06515392
Title: The Role of TIA Scores and NIHSS Score in Predicting Early and Late Ischemic Stroke Risk in Patients Presenting With Transient Ischemic Attack to the Emergency Department
Brief Title: TIA Scores' Mortality Predictions and Recurrent TIA and Stroke Prediction
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TIA Scores and Mortality
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic; Transient Ischemic Attack
Keywords: transient ischemic attack; ischemic stroke; TIA scores
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIA group: patients presenting with transient ischemic attack will be recorded and TIA scores and NIHSS score will be calculated, after 30 days follow-up, recurrent TIA and stroke rates will be determined

SUMMARY:
Our study adopts a prospective design. Our research aims to determine the significance of ABCD2, ABCD3-I, Canadian TIA Score, and NIHSS Score in predicting the likelihood of ischemic stroke within 30 days in patients presenting to the emergency department with transient ischemic attack (TIA)

DETAILED DESCRIPTION:
Our study is planned as follows: Patients diagnosed with transient ischemic attack (TIA) presenting to the emergency department will undergo scoring by researchers, although they will not intervene the treatment process of the patients. Patients will be contacted by researchers or their families to ascertain whether they experience a recurrent stroke or TIA within 30 days, and their current health status will be assessed. The collected information will be recorded.

The study will include patients diagnosed with transient ischemic attack (TIA) based on tests and imaging conducted at Ankara Etlik City Hospital's emergency department. The planned duration for data collection and analysis is one year.

Parameters to be examined:

Age Gender Physical examination findings Comorbidities (hypertension, coronary artery disease, valvular heart disease, COPD, asthma, diabetes, others) Neurological examination findings Time of symptom onset Admission status (intensive care unit / ward) Findings from ultrasound, computed tomography, and MRI imaging Length of hospital stay Mortality (yes/no)

We aim to collect data from approximately 300 patients within the course of one year for our study

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to the emergency department and diagnosed with TIA Patients diagnosed with ischemic stroke who did not receive thrombolytic therapy based on NIHSS score Patients aged 18 and above Patients who consented by signing the informed consent form

Exclusion Criteria:

Patients diagnosed with hemorrhagic stroke Patients unwilling to participate in the study Patients with a history of trauma Patients unable to receive thrombolytic therapy for any reason (trauma, malignancy, etc.) Patients under the age of 18 Patients transferred from another hospital Patients who experienced cardiac arrest Patients who died for any reason other than ischemic stroke within 30 days Patients wishing to withdraw from the study at any time during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 presenting to emergency department with symptoms of stroke and diagnosed with TIA will be enrolled to study and will be followed up for 30 days for recurrent TIA or stroke
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
recurrent TIA or stroke | 30 days
  recurrent TIA within 30 days of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perry JJ, Losier JH, Stiell IG, Sharma M, Abdulaziz K. National survey of emergency physicians for transient ischemic attack (TIA) risk stratification consensus and appropriate treatment for a given level of risk. CJEM. 2016 Jan;18(1):10-8. doi: 10.1017/cem.2015.57. Epub 2015 Jul 31. PMID 26226855
- [Background] Cortel-LeBlanc MA, Sharma M, Cortel-LeBlanc A, Sivilotti MLA, Emond M, Stiell IG, Stotts G, Lee J, Worster A, Morris J, Cheung KW, Jin AY, Oczkowski WJ, Sahlas DJ, Murray HE, Mackey A, Verreault S, Camden MC, Yip S, Teal P, Gladstone DJ, Boulos MI, Chagnon N, Shouldice E, Atzema C, Slaoui T, Teitelbaum J, Abdulaziz KE, Wells GA, Taljaard M, Perry JJ. Predictors of neurologists confirming or overturning emergency physicians' diagnosis of TIA or stroke. CJEM. 2021 Nov;23(6):812-819. doi: 10.1007/s43678-021-00181-0. Epub 2021 Sep 1. PMID 34468970
- [Background] Yang C, Jin A, Lin J, Wang Y, Xu J, Meng X. Validation of the Canadian TIA Score to Predict Subsequent Stroke Risk in Chinese TIA Patients. Cerebrovasc Dis. 2022;51(6):735-743. doi: 10.1159/000524264. Epub 2022 May 5. PMID 35512630